CLINICAL TRIAL: NCT06884033
Title: GINEMOTION: Cinematherapy for Women With Depression and Anxiety
Brief Title: Cinematherapy for Women With Depression and Anxiety
Acronym: GINEMOTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7075
Record Dates: First submitted 2025-03-10; First posted 2025-03-19 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-03

CONDITIONS: Depression Anxiety Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cinematherapy intervention (Experimental): Cinematherapy intervention
  Interventions: Behavioral: Cinematherapy

INTERVENTIONS:
Behavioral: Cinematherapy — Cinematherapy, also known as cinema therapy and movie therapy, involves therapist-directed viewing of movies for specific therapeutic purposes.

SUMMARY:
Group cinematherapy program in reducing depressive and anxiety symptoms in women diagnosed with Depressive Disorders and Anxiety Disorders.

DETAILED DESCRIPTION:
Cinematherapy is a creative therapeutic intervention in which a trained professional prescribes the patient to watch a film and uses the characters and themes as metaphors to promote self-exploration and change. The effectiveness of cinematherapy as a therapeutic technique has been demonstrated through its effectiveness in improving participants' self-esteem, emotional expression and understanding, and interpersonal relationships, and in reducing depressive and anxious symptoms.The cinematherapy intervention involves a targeted selection of film content and activities designed to improve the patients' mental condition.The study includes eight meetings on a monthly basis (programming of eight films lasting approximately two hours and subsequent discussion on the contents of the film shown).

ELIGIBILITY:
Inclusion Criteria:

* female, aged 18-75 years;
* Diagnosis of Depressive Disorders (unipolar and bipolar) and Anxiety Disorders according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5), both new onset in subjects without a previous psychiatric history, and depressive and anxious recurrences;
* Taking psychopharmacological therapy;
* Fluent knowledge of the Italian language;
* Release of a written informed consent, signed by the patient or legal representative and partner.

Exclusion Criteria:

* Diagnosis of Schizophrenia or other psychotic spectrum disorders;
* Diagnosis of neurological disorders associated with cognitive decline;
* Current abuse of alcohol and psychotropic substances, with the exception of smoking;
* Refusal to sign the informed consent to participate in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Assessment of change from baseline in anxiety symptoms. | 8 months
  The presence and degree of anxiety will be assessed using the Hamilton Anxiety Rating Scale (HARS). The scale consists of 14 items designed to assess the severity of a patient's anxiety. Each of the 14 items contains a number of symptoms, and each group of symptoms is rated on a scale of zero to four, with four being the most severe. A score of 17 or less indicates mild anxiety severity. A score from 18 to 24 indicates mild to moderate anxiety severity. Lastly, a score of 25 to 30 indicates a moderate to severe anxiety severity.
Assessment of change from baseline in depression symptoms. | 8 months
  The presence and degree of depression will be assessed using the Hamilton Depression Rating Scale (HDRS). The scale contains 17 items pertaining to symptoms of depression experienced over the past week. A score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher (indicating at least moderate severity) is usually required for entry into a clinical trial.

SECONDARY OUTCOMES:
Weight will be collected for all patients. | 8 months
  Weight in kilograms will be collected for all patients.
Eight will be collected for all patients. | 8 months
  Height in metres will be collected for all patients.
Body mass index (BMI) will be collected for all patients. | 8 months
  Body mass index, or BMI, gives an indication of body size. BMI is calculated using weight and height (weight in kilograms divided by height in metres squared).The formula is BMI = kg/m2; kg is a person's weight in kilograms and m2 is height in metres squared. BMI can help estimate risk of a heart attack or stroke.
Heart rate variability (HRV) will be collected for all patients. | 8 months
  HRV is a measure of the variation in time between each heartbeat in electrocardiogram . It is used as a reliable, noninvasive method of measuring physiological responses to stress. A consistent baseline score of 70 or higher is associated with health; whereas levels between 50 and 70 are compromised health and diseases; whereas a regular HRV below 50 puts the person at risk for catastrophic illness and even death.

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Mazza, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Marianna Mazza, Rome, ROMA, Italy

IPD SHARING:
Plan to Share IPD: No